CLINICAL TRIAL: NCT03384394
Title: Evaluating High-flow Nasal Cannula Oxygen Therapy Through Lung Ultrasound Score
Brief Title: Evaluating High-flow Nasal Cannula Oxygen Therapy Through LUS During Weaning
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: lu xiao (Other)
Responsible Party: Sponsor-Investigator, lu xiao, Principal Investigator,Second Affiliated Hospital, School of Medicine, Zhejiang University, Second Affiliated Hospital, School of Medicine, Zhejiang University
Organization: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 214856056
Record Dates: First submitted 2017-05-01; First posted 2017-12-27 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: High-flow Nasal Cannula Oxygen

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional oxygen therapy (Placebo Comparator): oxygen by a standard nasal cannula or nonrebreather mask
  Interventions: Device: Conventional oxygen therapy
- High-flow Nasal Cannula Oxygen Therapy (Active Comparator): High-flow Nasal Cannula Oxygen Therapy
  Interventions: Device: high-flow nasal cannula oxygen

INTERVENTIONS:
Device: high-flow nasal cannula oxygen — high-flow nasal cannula oxygen
  Arms: High-flow Nasal Cannula Oxygen Therapy
Device: Conventional oxygen therapy — oxygen by a standard nasal cannula or nonrebreather mask
  Arms: Conventional oxygen therapy

SUMMARY:
Respiratory distress after extubation is associated with increased morbidity and mortality. Its multifactorial pathophysiology causes a loss of pulmonary aeration during the weaning process, the clinical translation being impaired gas exchange and the occurrence of respiratory distress. Lung ultrasound can accurately quantify the loss of pulmonary aeration before, after end during the weaning trial by calculating the Lung Ultrasound Score (LUS). Investigators have recently demonstrated in a prospective two-center study of 100 patients that the intensity of the lung aeration loss occurring during the weaning trial, was predictive of the development of postextubation respiratory distress within 48 hours following extubation. A LUS ≥ 14 could identify patients at high risk of developing postextubation respiratory distress. A second study that investigators have just completed in 80 patients weaned from mechanical ventilation shows a 30% reduction of respiratory distress in post-extubation High Flow Nasal Cannula oxygen group compared to a standard O2 group.

The establishment of a targeted therapeutic strategy proposed in a group of high-risk patients, defined as having a ≥ 14 LUS at the end of the weaning trial could reduce the incidence of extubation failure and associated morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* patients above 18, mechanically ventilated on tracheal intubation for more than 48 hours.

Exclusion Criteria:

* Patients with chronic obstructive pulmonary disease (COPD) with moderate to severe (3 and 4) stage defined by a forced expiratory volume in one second (FEV) <50% of theoretical value
* Patients with previous chronic respiratory disease
* Paraplegia with level> T8,
* Severe ICU-acquired neuromyopathy
* Patients with tracheostomy for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2018-03-01 (Estimated); Primary Completion 2019-06-15 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
To decrease the incidence of extubation failure within 48 hours after a successful spontaneous breathing trial in ICU patients. | 48 hours
  To decrease the incidence of extubation failure within 48 hours after a successful spontaneous breathing trial in ICU patients.

SECONDARY OUTCOMES:
Number of ventilation-free days in ICU following the planned extubation after randomization. - Length of stay in ICU and in-hospital after randomization. - Mortality in ICU and at three months. | treatment in ICU and at three months.
  Number of ventilation-free days and mortality in ICU and at three months.

IPD SHARING:
Plan to Share IPD: Undecided